CLINICAL TRIAL: NCT06717529
Title: Functional and Clinical Outcomes of Hyaluronic Acid and Steroid Injections in Bilateral Knee Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Edin Mešanović (Other)
Responsible Party: Sponsor-Investigator, Edin Mešanović, Orthopedic surgeon, Cantonal Hospital Dr. Safet Mujic Mostar
Organization: Cantonal Hospital Dr. Safet Mujic Mostar (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01-1-1-5469/23-01
Record Dates: First submitted 2024-11-30; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Osteoarthritis (OA) of the Knee; Osteoarthritis; Osteoarthritis in the Knee; Osteoarthritis of Knee; Osteoarthritis of the Knees; Osteoarthritis of Knee Joint; Osteoarthritis Knee; Osteoarthritis of the Knee
Keywords: osteoarthritis; hyaluronic acid; steroid injection; kellgren lawrence; oa; arthritis
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee; Arthritis | interventions — Hyaluronic Acid; Methylprednisolone Acetate

STUDY DESIGN:
Intervention Model Description: Patients with bilateral knee osteoarthritis will receive hyaluronic acid injection in one knee and steroid injection in the other knee.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyaluronic acid injection (Experimental): This arm will receive a hyaluronic acid injection in the knee joint.
  Interventions: Other: Sodium hyaluronate (hyaluronic acid)
- Steroid injection (Active Comparator): This arm will receive steroid injection in the knee joint.
  Interventions: Drug: Methylprednisolone Acetate Injection

INTERVENTIONS:
Other: Sodium hyaluronate (hyaluronic acid) — The patient will receive one 3mL Sodium Hyaluronate injection containing 75 mg of active substance in one knee joint.
  Arms: Hyaluronic acid injection
Drug: Methylprednisolone Acetate Injection — The patient will receive 2mL of methylprednisolone acetate solution containing 80 mg of the medicine in other knee joint.
  Arms: Steroid injection

SUMMARY:
The aim of this study is to compare functional and clinical outcomes of intraarticular injections of hyaluronic acid and steroids in patients with bilateral knee osteoarthritis. We will compare clinical and functional outcomes for each knee separately after week 6, month 3, month 6, and one year after the intervention.

DETAILED DESCRIPTION:
We will include patients with bilateral knee osteoarthritis (Kellgren Lawrence grades 2 and 3). On initial examination, we will measure active and passive range of flexion and extension, presence of swelling, joint effusion, VAS score for each knee separately, and WOMAC score for every knee separately. We will randomly apply hyaluronic acid injection in one knee and steroid injection in the other knee. We will repeat the same examination after week 6, month 3, month 6, and one year after the procedure. The main aim is to check whether there is a significant clinical or functional difference between two groups.

ELIGIBILITY:
Inclusion Criteria:

* bilateral knee pain
* same grade of osteoarthritis in both knees
* Kellgren-Lawrence grade 2 or 3 of knee osteoarthritis
* fully completed all follow-up examinations

Exclusion Criteria:

* unilateral knee osteoarthritis
* different grade of osteoarthritis between knees based on Kellgren-Lawrence scale
* positive history of previous knee interventions (injections, surgery)
* positive history of additional knee injuries (meniscus, ligament...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
WOMAC score | One year after the intervention.
  Changes in WOMAC score one year after the intervention compared to the WOMAC score at the initial examination.
VAS score | One year after the intervention.
  Changes in VAS score after one year.
Range of active knee joint flexion | One year after the intervention.
  Changes in the range of active knee joint flexion
Range of active knee joint extension | One year after the intervention.
  Changes in the range of active knee joint extension
Knee swelling | One year after the intervention.
  Presence of knee joint swelling.
Knee joint effusion | One year after the intervention.
  The presence of knee joint effusion.

SECONDARY OUTCOMES:
WOMAC score after 6 weeks | 6 weeks after the intervention.
  Changes in WOMAC score compared to the initial examination.
VAS score after 6 weeks | 6 weeks after the intervention.
  Changes in VAS score compared to the initial examination.
Range of active knee joint flexion after 6 weeks | 6 weeks after the intervention.
  Changes in range of active knee joint flexion compared to the initial examination.
Range of active knee joint extension after 6 weeks | 6 weeks after the intervention.
  Changes in the range of knee joint extension compared to the initial examination.
Knee swelling after 6 weeks | 6 weeks after the intervention.
  Changes in the presence of knee swelling compared to the initial examination.
Knee joint effusion after 6 weeks | 6 weeks after the intervention.
  Changes in the presence of knee joint effusion compared to the initial examination.
WOMAC score after 3 months | 3 months after the intervention.
  Changes in WOMAC score compared to the initial examination.
VAS score after 3 months | 3 months after the intervention.
  Changes in VAS score compared to the initial examination.
Range of active knee joint flexion after 3 months | 3 months after the intervention.
  Changes in the range of knee joint flexion compared to the initial examination.
Range of active knee joint extension after 3 months | 3 months after the intervention.
  Changes in the range of knee joint extension compared to the initial examination.
Knee swelling after 3 months | 3 months after the intervention.
  Changes in the presence of knee swelling compared to the initial examination.
Knee joint effusion after 3 months | 3 months after the intervention.
  Changes in the presence of knee joint effusion compared to the initial examination.
WOMAC score after 6 months | 6 months after the intervention.
  Changes in WOMAC score compared to the initial examination.
VAS score after 6 months | 6 months after the intervention.
  Changes in VAS score compared to the initial examination.
Range of active knee joint flexion after 6 months | 6 months after the intervention.
  Changes in the range of knee joint flexion compared to the initial examination.
Range of active knee joint extension after 6 months | 6 months after the intervention.
  Changes in the range of knee joint extension compared to the initial examination.
Knee swelling after 6 months | 6 months after the intervention.
  Changes in the presence of knee swelling compared to the initial examination.
Knee joint effusion after 6 months | 6 months after the intervention.
  Changes in the presence of knee effusion compared to the initial examination.

CONTACTS AND LOCATIONS:
Locations (1):
- Cantonal Hospital "dr.Safet Mujic", Mostar, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Ko NY, Chang CN, Cheng CH, Yu HK, Hu GC. Comparative Effectiveness of Focused Extracorporeal versus Radial Extracorporeal Shockwave Therapy for Knee Osteoarthritis-Randomized Controlled Study. Int J Environ Res Public Health. 2022 Jul 24;19(15):9001. doi: 10.3390/ijerph19159001. PMID 35897371
- [Background] Mitra, S., Seenappa, H., & Madhavan, P. (2021). A clinical evaluation study of single spin vs double spin intra-articular prp injection in patients with bilateral early oa knee: a novel technique. International Journal of Orthopaedics Sciences, 7(3), 01-06. https://doi.org/10.22271/ortho.2021.v7.i3a.2718
- [Background] Rahman, S., Narhari, P., Sharifudin, M., & Aa, S. (2020). Western ontario and mcmaster universities (womac) osteoarthritis index as an assessment tool to indicate total knee arthroplasty in patients with primary knee osteoarthritis. Iium Medical Journal Malaysia, 19(3). https://doi.org/10.31436/imjm.v19i3.1664
- [Background] Wang SZ, Wu DY, Chang Q, Guo YD, Wang C, Fan WM. Intra-articular, single-shot co-injection of hyaluronic acid and corticosteroids in knee osteoarthritis: A randomized controlled trial. Exp Ther Med. 2018 Sep;16(3):1928-1934. doi: 10.3892/etm.2018.6371. Epub 2018 Jun 29. PMID 30186420
- [Background] Metcalfe AJ, Andersson ML, Goodfellow R, Thorstensson CA. Is knee osteoarthritis a symmetrical disease? Analysis of a 12 year prospective cohort study. BMC Musculoskelet Disord. 2012 Aug 22;13:153. doi: 10.1186/1471-2474-13-153. PMID 22917179
- [Background] Khalaj N, Abu Osman NA, Mokhtar AH, George J, Abas WA. Effect of intra-articular hyaluronic injection on postural stability and risk of fall in patients with bilateral knee osteoarthritis. ScientificWorldJournal. 2014;2014:815184. doi: 10.1155/2014/815184. Epub 2014 Jun 19. PMID 25136689
- [Background] Cotofana S, Wirth W, Pena Rossi C, Eckstein F, Gunther OH. Contralateral knee effect on self-reported knee-specific function and global functional assessment: data from the Osteoarthritis Initiative. Arthritis Care Res (Hoboken). 2015 Mar;67(3):374-81. doi: 10.1002/acr.22495. PMID 25302424